CLINICAL TRIAL: NCT04937829
Title: Randomized, Double-blind (Patient, Investigator), Placebo-controlled, Parallel Group, Single Dosing Study on Safety, Tolerability, Pharmacokinetic and Preliminary Efficacy of BI 1569912 as Adjunctive Therapy in Patients With Major Depressive Disorder
Brief Title: A Study to Test How Well Different Doses of BI 1569912 Are Tolerated and How Well They Work in People With Depression Who Take Anti-depressive Medication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1447-0003
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1569912 treatment group (Experimental)
  Interventions: Drug: BI 1569912
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1569912 — BI 1569912
  Arms: BI 1569912 treatment group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This study is open to adults between 18 and 65 years of age who have depression (major depressive disorder). People with a current depressive episode lasting between 2 months and one and a half years can join the study. This study is for people for whom existing treatments for depression do not work sufficiently.

The purpose of this study is to test how well a medicine called BI 1569912 is tolerated and whether it may help people with depression.

It is planned to test 4 different dosages of BI 1569912 in this study. Each participant gets either one BI 1569912 dosage or placebo. It is decided randomly, which means by chance, who gets which treatment. Participants take BI 1569912 or placebo as tablets once during the study. Placebo tablets look like BI 1569912 tablets but do not contain any medicine. Participants also continue taking their usual medicine for depression throughout the study.

Participants are in the study for about 5 weeks. During this time, they visit the study site 4 times, with a stay at the study site for 9 days.

The doctors check the health of the participants and note any health problems that could have been caused by BI 1569912. The participants fill in questionnaires about their depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of Major Depressive Disorder (MDD) as confirmed at the time of screening by the Mini International Neuropsychiatric Interview (MINI), with a duration of current depressive episode ≥ 8 weeks and ≤ 24 months at the time of screening visit.
2. At least moderate severity of MDD confirmed by a trained site-based rater, at screening and Visit 2 day 1 (i.e. prior to randomisation). For patients who are not on an SSRI at Visit 1, MDD must be confirmed additionally at Visit 1 A.
3. In the current episode, patients have shown insufficient treatment response (defined by less than 50 % response to one or more antidepressant drugs of adequate dose and treatment duration (according to Summary of Product Characteristics) as evaluated by Antidepressant Treatment Response Questionnaire (ATRQ). Participants, who, in addition to their monotherapy with an SSRI/SNRI, are taking additional low dose antidepressant medications for purposes other than treating depressive symptoms, are not excluded. The dose must be less than the lowest dose indicated for MDD. Use of bupropion is not allowed.
4. Documented ongoing monotherapy treatment of ≥ 6 weeks at randomisation (i.e. Visit 2 day 1) with a protocol specified Selective Serotonin Reuptake Inhibitors (SSRI) or Serotonin-Norepinephrine Reuptake Inhibitors (SNRI) at adequate dose (according to ATRQ assessment). sampling at Visit 1). Patients who are not on an SSRI at Visit 1 will undergo a lead in phase as described in the Flow Chart. Patients who meet all the eligibility criteria but are not on an SSRI/SNRI at Visit 1, will have the option to undergo a 6 week open label lead in phase with SSRI/SNRI. These patients will be reassessed at Visit 1A to determine eligibility to be randomized to the trial.
5. Male or female patients, aged 18 to 65 years at screening. If Women of childbearing potential (WOCBP) are included, they have to be able and willing to use two methods of contraception which include one highly effective method of birth control per ICH M3 (R2) that result in a low failure rate of less than 1 %, plus one additional barrier method. If men who are able to father a child, are willing to participate, they have to use an adequate form of effective contraception for the duration of study participation and for at least 28 days after treatment has ended.
6. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial. Please note complete sexual abstinence is allowed when this is in line with the preferred and usual lifestyle of the patient (note: periodic abstinence such as calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception) - (in this specific case the barrier methods, as mentioned below, are not applicable). Sexual abstinence as a contraceptive method will not be allowed for WOCBP who are heterosexually active.

Exclusion Criteria:

1. Patient had met diagnostic criteria per Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, delusional disorder or MDD with psychotic features at any time point in the patient's life.
2. Diagnosis with antisocial, paranoid, schizoid, schizotypical or Borderline personality disorder as per DSM-5 criteria at the time of screening visit. Any other personality disorder at screening visit that significantly affects current psychiatric status and is likely to impact trial participation, as per the judgement of investigator.
3. Diagnosis of any other mental disorder (in addition to those as described in Exclusion Criterion #1 and #2) that was the primary focus of treatment within 6 months prior to screening, as per clinical discretion of the investigator.
4. Patients with a Body Mass Index (weight [kg]/height [m]²) lower than 18 kg/m² at screening.
5. Diagnosis of a moderate to severe substance-related disorder within the last 6 months before screening visit (with exception of caffeine and tobacco).
6. Use of Ketamine/S-Ketamine for the current ongoing depressive episode.
7. Stable treatment with benzodiazepines and/or nonbenzodiazepine hypnotics. (Note: As needed (PRN) use of benzodiazepines and/or nonbenzodiazepine hypnotics may be acceptable except for the trial period Day -1 to Day 2).

Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with drug-related adverse events (AEs) | Up to Day 15
Maximum decrease from baseline (peak decrease) in Montgomery-Åsberg Depression Rating Scale (MADRS) at any day within a 7 days-interval | Up to Day 15
  MADRS is a ten-item questionnaire used to measure the severity of Major Depressive Disorder (MDD). Nine of the items are based upon patient reports and one is on the rater's observation (apparent sadness) during the rating interview. MADRS items are rated on a 0 to 6 continuum (0=no abnormality, 6=severe). The possible total score could range from 0 to 60 (from normal with absence of symptoms to severe depression).

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale Area under the response curve from pre-dose to the last measurement during inpatient stay at 166:30 hours (MADRS AUC0-166:30) | Up to Day 15
  MADRS is a ten-item questionnaire used to measure the severity of Major Depressive Disorder (MDD). Nine of the items are based upon patient reports and one is on the rater's observation (apparent sadness) during the rating interview. MADRS items are rated on a 0 to 6 continuum (0=no abnormality, 6=severe). The possible total score could range from 0 to 60 (from normal with absence of symptoms to severe depression).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Collaborative Neuroscience Network, LLC (CNS), Garden Grove, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Optimus U Corporation, Miami, Florida
  - Research Centers of America, Oakland Park, Florida
  - iResearch Atlanta, Decatur, Georgia
  - Hassman Research Institute, Berlin, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - InSite Clinical Research, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com